CLINICAL TRIAL: NCT04985734
Title: Study on the Occurrence of Transthyretin Amyloidosis Cardiomyopathy in Patients With Idiopathic Peripheral Neuropathy
Brief Title: Transthyretin Amyloidosis Cardiomyopathy (ATTR-CM) in Patients With Idiopathic Peripheral Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: EDGE1850
Record Dates: First submitted 2021-05-17; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Amyloidosis Cardiac; Amyloid Polyneuropathy; Amyloidosis; Heart Failure; Cardiomyopathy Non-Dilated; Cardiomyopathies, Secondary
Keywords: Amyloidosis Cardiac; Amyloid Polyneuropathy; Amyloidosis; Heart Failure; Cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Amyloid Neuropathies; Amyloidosis; Heart Failure; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: Cohort of patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients under diagnostic work-up (Experimental)
  Interventions: Diagnostic Test: Specific diagnostic work-up for ATTR-CM patients

INTERVENTIONS:
Diagnostic Test: Specific diagnostic work-up for ATTR-CM patients — Technetium-scintigraphy

SUMMARY:
The goal of the present study is to determine the occurrence of wild-type and hereditary transthyretin amyloidosis cardiomyopathy among patients with the diagnosis of idiopathic peripheral neuropathy in the setting of a state-of-the-art diagnostic work-up; the investigators believe that the identification of patients with ATTR-CM in this setting can contribute to the early diagnosis of a largely underrecognized condition and, therefore, offer conditions to timely initiation of appropriate therapy with impact on prognosis of patients.

DETAILED DESCRIPTION:
Background. Different studies have described the value of amyloidosis screening in different clinical settings. The investigators hypothesize that in a relevant yet undetermined proportion of patients with idiopathic peripheral neuropathy a concomitant diagnosis of transthyretin amyloidosis cardiomyopathy can be made with a modern diagnostic work-up based on Technetium-scintigraphy as the primary screening tool. Further the investigators believe that the identification of these patients can lead to early initiation of therapy and modification of the prognosis of the disease.

Objective. To study the occurrence of transthyretin amyloidosis cardiomyopathy in patients with a diagnosis of idiopathic peripheral neuropathy using Tc-scinfigraphy as the primary screening tool.

Methods. This will be a prospective longitudinal cohort of adult patients with the diagnosis of idiopathic peripheral neuropathy. All patients will be submitted to a cardiologic evaluation that will include clinical evaluation, laboratory tests, electrocardiogram and echocardiography. For the diagnosis of amyloidosis all patients will be submitted to 99mTc-Methyl-Diphosphonate scintigraphy. Those with a positive result (grade 2 to 3 cardiac uptake) will be considered as having diagnosis of transthyretin amyloidosis cardiomyopathy and will be further submitted to genetic testing for transthyretin mutation; patients with abnormal scintigraphic results that do not meet current semi-quantitative diagnostic criteria will be submitted to additional investigation, that will include magnetic resonance heart imaging and fat biopsy. All patients will receive standard care for heart failure and transthyretin amyloidosis cardiomyopathy and will be follow-up every 6 months with clinical parameters, quality life questionnaire, ergospirometer and echocardiogram Perspectives. The investigators believe that the identification of patients with transthyretin amyloidosis cardiomyopathy in this setting can contribute to the early diagnosis of a largely underrecognized condition and, therefore, offer conditions to timely initiate appropriate therapy with impact on prognosis of patients.

ELIGIBILITY:
Inclusion Criteria

- Adult patients (> 18 years old) with diagnosis of idiopathic peripheral neuropathy

Exclusion criteria

* Patients with alternative established diagnosis of heart disease (ischemic heart disease, primary valvular heart disease, cardiomyopathies, pericardial disease)
* Patients with end stage renal disease undergoing dialysis
* Patients with other medical conditions recognized to impair the 1-year prognosis of patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis yield | 1 year
  Diagnosis yield of Tc-scintigraphy as a screening tool for ATTR-CM, as measured by the percentage of patients with a confirmed diagnosis of ATTR-CM in relation to the whole population of patients studied

CONTACTS AND LOCATIONS:
Locations (1):
- Emeline van Craenenbroek, Edegem, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: Undecided